CLINICAL TRIAL: NCT04751656
Title: Preventing Weight Gain Among Those Who Decline Behavioral Weight Loss Treatment
Brief Title: Preventing Weight Gain Among Those Who Decline Behavioral Weight Loss Treatment (STEADY)
Acronym: STEADY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB202001935-N-R; 5R03HL154272-02 (NIH); AWD08696 (Other: UFIRST Awards)
Record Dates: First submitted 2021-02-09; First posted 2021-02-12 (Actual); Results first posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-12

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Single-arm trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Steady Intervention (Experimental): Participants asked to engage in Steady Intervention for 12 months
  Interventions: Behavioral: Steady Intervention

INTERVENTIONS:
Behavioral: Steady Intervention — Participants will be asked to weigh themselves daily via a "smart" scale that transmits weight data directly to the study team via the cellular network for 12 months. Every-other week, participants will be sent text messages providing brief feedback encouraging continued self-weighing. Moreover, if a small weight gain is observed, participants will be sent text messages aiming to engage them in commercial or community-based evidence-based weight management resources.

SUMMARY:
The goal of this pilot trial is to pilot test an intervention to help prevent weight gain or produce weight loss among adults with obesity. Participants are asked to self-weigh on a smart scale for one year. Feasibility and acceptability outcomes are examined.

DETAILED DESCRIPTION:
To prevent weight gain while overcoming these common barriers to engaging in weight management interventions, we propose an intervention that prescribes self-weighing but does not prescribe changes in diet or physical activity behaviors or require attendance at didactic-focused meetings. The potential of self-weighing to promote weight management is supported both by self-regulatory theory and empirical research. Promoting self-weighing may activate participants' self-regulatory skills, leading to spontaneous decisions to reduce calorie intake or increase physical activity, thus preventing further weight gain. The proposed intervention will also provide individuals with text message-based feedback to promote continued self-weighing and to motivate engagement with evidence-based resources for weight management at a time when they may be more open to using these resources-e.g., after experiencing a small weight gain. The current proposal will investigate the feasibility and acceptability of this low burden self-weighing intervention in order to prepare for a fully-powered, pragmatic randomized controlled trial. We will enroll 40 patients with either obesity or overweight with a weight-related comorbidity and who have declined to participate in a comprehensive behavioral weight management program. Participants will be asked to weigh themselves daily via a "smart" scale that transmits weight data directly to the study team via the cellular network. Every-other week, participants will be sent text messages providing brief feedback encouraging continued self-weighing. Moreover, if a small weight gain is observed, participants will be sent text messages aiming to engage them in commercial or community-based evidence-based weight management resources. In a single-arm design, all enrolled participants will receive the intervention for 12 months and will complete assessments at 3 and 12 months to assess feasibility and acceptability of the intervention and trial design, while weight will be obtained from participants' Electronic Health Records (EHR). We will evaluate our success in meeting pre-specified metrics for trial feasibility and intervention acceptability outcomes, including intervention enrollment, intervention satisfaction, and obtainment of weight data abstracted from participants' EHRs. We will also evaluate the success of the intervention in promoting regular self-weighing and use of evidence-based weight management resources.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* Body weight recorded in EHR in the prior month from a primary care setting.
* Last BMI in EHR either ≥30 kg/m2 or between 25.0-29.9 kg/m2 with documented weight-related comorbidity (hypertension, type II diabetes, pre-diabetes, dyslipidemia, sleep apnea).
* Weight ≤ 375 lbs.
* Self-report sending and receiving at least one text message per month for past 6 months.
* Not currently enrolled in comprehensive behavioral weight loss treatment.
* Respond "no" to question asking if they would like to enroll in a comprehensive weight loss program in the next month
* Has not engaged in self-weighing ≥ 5 times per week on average over prior month.
* Not pregnant, breastfeeding, or planning to become pregnant in next 6 months.
* Not currently undergoing radiation or chemotherapy for cancer.
* No history of eating disorders.
* Interested in enrolling in low-burden self-weighing intervention.
* Able to read and understand English without help

Exclusion criteria:

* History of Congestive Heart Failure or heart attack in past 6 months.
* Planning to move out of the region in the following 12 months
* Answer incorrectly on an attention check/ validation survey item

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan McVay, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Health at the University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
The dataset will be prepared according to requirements for NHLBI data repository datasets and will be stored in the NHLBI data repository.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Per guidelines for sharing in the NHLBI repository, the data set will be submitted to the NHLBI program officer as soon as it is prepared, and no later than 3 years after the end of clinical activities.
Access Criteria: Consistent with NHLBI repository guidelines.

RESULTS

PARTICIPANT FLOW:
Groups:
- Steady Intervention Enrollees: Participants who enrolled in the Steady Intervention
Period: Overall Study
Arm/Group | Steady Intervention Enrollees
Started | 39
Completed | 38
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Steady Intervention Enrollees
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 24
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Intervention Satisfaction
Description: (NOTE: this is a pilot study and there is not a true primary outcome. There are several descriptive outcomes that will inform our decision to proceed to a traditional, fully powered clincial trial).
  Intervention satisfaction reported here is response to item "overall, I am satisfied with this program." with response options 1-5, 1-strongly disagree, 3-neither agree nor disagree, and 5-strongly agree.
Time Frame: 12 months.
Population: Those who completed 12 month assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steady Intervention Enrollees
Number analyzed (Participants) | 34
score on a scale | 4.1 (1.0)

2. Secondary Outcome: Retention in Study
Description: Percent of participants completing 12 month survey. (There is no measurement used for this. It is based on the portion of patients who complete the 12 month survey.)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Steady Intervention Enrollees
Number analyzed (Participants) | 39
Participants | 34

3. Secondary Outcome: Engagement in Self Weighing, First Quarter
Description: days/week in which weight was registered
Time Frame: months 0-3
Measure: Mean (Standard Deviation); unit: days/week
Arm/Group | Steady Intervention Enrollees
Number analyzed (Participants) | 39
days/week | 4.9 (1.2)

4. Secondary Outcome: Engagement in Self Weighing, Final Quarter
Description: mean days per week in which weight was registered
Time Frame: months 9-12
Measure: Mean (Standard Deviation); unit: days/week
Arm/Group | Steady Intervention Enrollees
Number analyzed (Participants) | 39
days/week | 4.2 (1.7)

5. Secondary Outcome: Percent of Patients Who Enroll
Description: Percent of those who are eligible who are interested in and enroll in the Steady Intervention out of those who complete the screening measure.
Time Frame: at recruitment
Population: those who were offered steady
Measure: Count of Participants; unit: Participants
Arm/Group | Steady Intervention
Number analyzed (Participants) | 86
Participants | 39

6. Secondary Outcome: Representatives of Those Who Enroll
Description: Percent of those participants who enroll who are male.
Time Frame: At recruitment
Measure: Count of Participants; unit: Participants
Arm/Group | Steady Intervention Enrollees
Number analyzed (Participants) | 39
Participants | 20

7. Secondary Outcome: Use of Evidence-based Resources Offered
Description: Percent of patients who initiate use of comprehensive weight loss program
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Steady Intervention Enrollees
Number analyzed (Participants) | 39
Participants | 3

ADVERSE EVENTS:
Time Frame: 1 year
Description: adverse events could be spontaneously reported to study staff. No formal assessment of adverse events was done.
Arm/Group | Steady Intervention Enrollees
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-04): https://cdn.clinicaltrials.gov/large-docs/56/NCT04751656/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/56/NCT04751656/ICF_001.pdf